CLINICAL TRIAL: NCT00467259
Title: A Randomized, Double-Blind, Placebo-controlled, Multicenter, 52-week Study to Evaluate the Endometrial Safety of Transdermal Testosterone (300 Mcg/Day) in Naturally Postmenopausal Women With Hypoactive Sexual Desire Disorder.
Brief Title: Endometrial Safety Study of Transdermal Testosterone (300 Mcg/Day) in Naturally Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007004
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-11

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Natural Menopause
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 28 cm² Placebo patch
  Interventions: Drug: Placebo patch
- Testosterone (Experimental): Testosterone patch, 300 mcg/day, change patch twice a week for 52 weeks
  Interventions: Drug: Testosterone Transdermal System

INTERVENTIONS:
Drug: Testosterone Transdermal System — Testosterone patch, 300 mcg/day, change patch twice a week for 52 weeks
  Arms: Testosterone
Drug: Placebo patch — placebo patch, changed twice a week for 52 weeks
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the endometrial safety of a testosterone patch as treatment for low libido in naturally postmenopausal women.

DETAILED DESCRIPTION:
Naturally postmenopausal women with hypoactive sexual desire disorder (HSDD) will be randomized into a 52-week, multicenter, double-blind (DB), parallel-group, placebo-controlled study. Patients will be stratified based on whether they use concomitant estrogen/progestin therapy and then randomized in a 4:1 ration to receive either testosterone transdermal system (300 mcg/day) or placebo. Patients using estrogen/progestin at the start of the study should maintain this therapy throughout the study; patients not using estrogen/progestin at the start of the study should not initiate estrogen/progestin therapy throughout the study. Endometrial biopsies and transvaginal ultrasounds will be collected/performed at screening and study exit for all patients. Safety will be assessed by adverse events, reports of vaginal bleeding, lipids, serum chemistry, and hematology. Physical exams, pap smears, and mammograms will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Women will be screened for study participation and must be at least one year post menopausal, 45-70 years old, in general good health, and may or may not be on hormone therapy, and must have low sexual desire which causes distress.

Exclusion Criteria:

* Women will be screened for study participation and must not be using androgen therapy or have any medical, physical, psychological, or pharmacological condition that could make participation unsafe or confound the safety evaluation.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1271 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johna Lucas, MD, Study Director — Procter and Gamble
Locations (111):
- United States (111):
  - Study Facility, Birmingham, Alabama
  - Research Facility, Birmingham, Alabama
  - Research Facility, Mobile, Alabama
  - Research Facility, Montgomery, Alabama
  - Test Facility, Chandler, Arizona
  - Study Facility, Peoria, Arizona
  - Research Facility, Phoenix, Arizona
  - Research Facility, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Facility, Tucson, Arizona
  - Study Facility, Tuscon, Arizona
  - Site Facility, Jonesboro, Arkansas
  - Site Facility, Little Rock, Arkansas
  - Research Facility, Anaheim, California
  - Research Site, Berkeley, California
  - Research Facility, Palm Desert, California
  - Research Facility, Pasadena, California
  - Research Facility, San Diego, California
  - Research Facility, San Ramon, California
  - Test Facility, Santa Rosa, California
  - Site Facility, Upland, California
  - Research Facility, Vista, California
  - Site Facility, Vista, California
  - Site Facility, Westlake Village, California
  - Test Facility, Denver, Colorado
  - Research Facility, Longmont, Colorado
  - Test Facility, New London, Connecticut
  - Study Facility, Waterbury, Connecticut
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Boynton Beach, Florida
  - Site Facility, Clearwater, Florida
  - Site Facility, Daytona Beach, Florida
  - Research Facility, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Site Facility, Jupiter, Florida
  - Test Facility, Miami, Florida
  - Research Facility, Pinellas Park, Florida
  - Research Facility, Plantation, Florida
  - Study Facility, South Miami, Florida
  - Research Site, Tampa, Florida
  - Test Facility, Vero Beach, Florida
  - Research Facility, West Palm Beach, Florida
  - Research Facility, Weston, Florida
  - Research Facility, Alpharetta, Georgia
  - Research Facility, Atlanta, Georgia
  - Site Facility, Decatur, Georgia
  - Site Facility, Douglasville, Georgia
  - Site Facility, Roswell, Georgia
  - Test Facility, Savannah, Georgia
  - Study Facility, Idaho Falls, Idaho
  - Test Facility, Champaign, Illinois
  - Test Facility, Chicago, Illinois
  - Test Facility, Indianapolis, Indiana
  - Research Facility, Overland Park, Kansas
  - Site Facility, Louisville, Kentucky
  - Study Facility, Baltimore, Maryland
  - Research Facility, Baltimore, Maryland
  - Study Facility, Boston, Massachusetts
  - Research Facility, Bingham Farm, Michigan
  - Study Facility, Paw Paw, Michigan
  - Test Facility, Saginaw, Michigan
  - Research Facility, Edina, Minnesota
  - Research Site, Jackson, Mississippi
  - Test Facility, St Louis, Missouri
  - Site Facility, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Site Facility, Las Vegas, Nevada
  - Test Facility, Reno, Nevada
  - Test Facility, Moorestown, New Jersey
  - Research Facility, New York, New York
  - Test Facility, Raleigh, North Carolina
  - Site Facility, Winston-Salem, North Carolina
  - Study Facility, Winston-Salem, North Carolina
  - Research Facility, Beachwood, Ohio
  - Test Facility, Centerville, Ohio
  - Research Facility, Cincinnati, Ohio
  - Study Facility, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Site Facility, Cleveland, Ohio
  - Test Facility, Columbus, Ohio
  - Research Facility, Dayton, Ohio
  - Test Facility, Englewood, Ohio
  - Test Facility, Oklahoma City, Oklahoma
  - Test Facility, Tulsa, Oklahoma
  - Site Facility, Eugene, Oregon
  - Research Facility, Philadelphia, Pennsylvania
  - Study Facility, Bristol, Tennessee
  - Research Facility, Chattanooga, Tennessee
  - Research Facility, Nashville, Tennessee
  - Site Facility, Austin, Texas
  - Research Facility, Carrolton, Texas
  - Site Facility, Corpus Christi, Texas
  - Research Facility, Dallas, Texas
  - Test Facility, Farmers Branch, Texas
  - Research Facility, Houston, Texas
  - Research Facility, Irving, Texas
  - Research Facility, Midland, Texas
  - Research Facility, Richardson, Texas
  - Site Facility, San Antonio, Texas
  - Test Facility, San Antonio, Texas
  - Study Facility, Salt Lake City, Utah
  - Research Facility, West Valley City, Utah
  - Research Facility, Newport News, Virginia
  - Study Facility, Richmond, Virginia
  - Test Facility, Richmond, Virginia
  - Site Facility, Richmond, Virginia
  - Research Facility, Virginia Beach, Virginia
  - Site Facility, Seattle, Washington
  - Research Facility, Tacoma, Washington
  - Test Facility, Tacoma, Washington
  - Research Site, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began 14 May 2007
Pre-assignment Details: Randomized 1127 women not using concomitant estrogen & progestin (E&P) therapy. An additional 134 women using concomitant estrogen & progestin therapy were randomized. Subjects were stratified by using or not using E&P by site and then randomized 4:1 300 mcg/d TTS or placebo.
Groups:
- Placebo: Placebo patch
Period: Overall Study
Arm/Group | Placebo | Testosterone
Started | 251 | 1020
ITT Population | 251 | 1019 (One subject did not take any study medication and was excluded from ITT population.)
Completed | 176 | 778
Not Completed | 75 | 242
Not completed — Adverse Event | 24 | 90
Not completed — Protocol Violation | 1 | 7
Not completed — Withdrawal by Subject | 34 | 108
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 14 | 34
Not completed — Site Closed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Testosterone | Total
Number analyzed (Participants) | 251 | 1020 | 1271
Age Continuous [Mean (Standard Deviation); unit: years] — ITT Population
  years | 55.5 (4.8) | 55.8 (4.9) | 55.7 (4.9)
Age, Customized [Number; unit: Participants] — ITT Population
  Participants
    40-49 years old | 21 | 95 | 116
    50-59 years old | 182 | 700 | 882
    60-65 years old | 39 | 189 | 228
    66 + years old | 9 | 35 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 1020 | 1271
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Number; unit: Participants] — ITT Population
  Participants
    Hispanic or Latino | 14 | 50 | 64
    Not Hispanic or Latino | 237 | 969 | 1206
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — ITT Population
  Participants
    Indian (American) | 1 | 3 | 4
    Asian (Oriental) | 3 | 6 | 9
    Black or African American | 9 | 82 | 91
    Caucasian | 231 | 920 | 1151
    Hispanic | 1 | 3 | 4
    Indian (Asian) | 0 | 1 | 1
    Latino | 0 | 2 | 2
    Mexican | 1 | 0 | 1
    Multi-Racial | 4 | 1 | 5
    Hawaiian / Pacific Islander | 0 | 1 | 1
    Spanish | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 251 | 1020 | 1271

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Endometrial Hyperplasia in Naturally Postmenopausal Women With Hypoactive Sexual Desire Disorder (HSDD) Not Using Concomitant Estrogen and Progestin, Year 1
Description: Incidence measured is number of patients with endometrial hyperplasia/number of patients with evaluable biopsies
Time Frame: 52 weeks
Population: Subjects with evaluable endometrial biopsies.
Measure: Number (95% Confidence Interval); unit: # Endometrial Hyperplasia/Evaluable Biop
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 137 | 580
# Endometrial Hyperplasia/Evaluable Biop | 0 [0 to 2.6] | 0 [0 to 0.6]
Statistical Analysis 1: Comparison: Placebo vs Testosterone; 1000 naturally postmenopausal women not on concomitant E+P therapy at baseline were to be randomized (800 TTS; 200 placebo). It was assumed 60% would complete 1 year and 80% of these would have evaluable biopsies. Of the 800 randomized to TTS approximately 380 were expected to have evaluable biopsies at 1 year. 380 patients on TTS with evaluable biopsies at 1 year would provide 90% power to rule out an incidence of hyperplasia of 2% using the upper bound of a 2-sided 95% CI; Test type: Superiority or Other; p = 1.0000, Fisher Exact; p-value obtained from Fisher's exact test and corresponds to the test of the null hypothesis of no treatment difference

2. Secondary Outcome: Incidence of Endometrial Hyperplasia in Naturally Postmenopausal Women With HSDD Using Concomitant Estrogen and Progestin, Year 1
Description: Incidence measured is number of patients with endometrial hyperplasia/number of patients with evaluable biopsies
Time Frame: 52 weeks
Population: Subjects with evaluable endometrial biopsies.
Measure: Number (95% Confidence Interval); unit: # Endometrial Hyperplasia/Evaluable Biop
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 10 | 68
# Endometrial Hyperplasia/Evaluable Biop | 0 [0 to 26.7] | 0 [0 to 5.2]
Statistical Analysis 1: Comparison: Placebo vs Testosterone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact; p-value obtained from Fisher's exact test and corresponds to the test of the null hypothesis of no treatment difference

3. Secondary Outcome: Incidence Endometrial Hyperplasia in Naturally Postmenopausal Women With HSDD Using Concomitant Estrogen & Progestin Combined With Those Not Using Estrogen & Progestin Therapy, Year 1
Description: Incidence measured is number of patients with endometrial hyperplasia/number of patients with evaluable biopsies
Time Frame: 52 weeks
Population: Subjects with evaluable endometrial biopsies.
Measure: Number (95% Confidence Interval); unit: # Endometrial Hyperplasia/Evaluable Biop
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 147 | 648
# Endometrial Hyperplasia/Evaluable Biop | 0 [0 to 2.4] | 0 [0 to 0.5]
Statistical Analysis 1: Comparison: Placebo vs Testosterone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact; p-value obtained from Fisher's Exact test and corresponds to the test of the null hypothesis of no treatment difference

ADVERSE EVENTS:
Time Frame: 52 week treatment period
Description: Vaginal bleeding that worsens from baseline will only be recorded on vaginal bleeding page, not as an AE. However, if vaginal bleeding results in study withdrawal or meets the ICH definition of a "serious" AE it will be recorded as an AE.
Arm/Group | Placebo | Testosterone
Serious Adverse Events (participants affected / at risk) | 10/251 | 33/1019
Other Adverse Events (participants affected / at risk) | 125/251 | 472/1019
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=251) | Testosterone (N=1019)
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Congenital Cerebrovascular Anomaly (Congenital, familial and genetic disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Oesophageal Spasm (Gastrointestinal disorders) | 1 | 0
Small Intestine Haemorrhage (Gastrointestinal disorders) | 1 | 0
Appendicitis Perforated (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Joint Abscess (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Sternal Injury (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthritis Reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1
Carotid Artery Occlusion (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 3
Affective Disorder (Psychiatric disorders) | 0 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Glomerulonephritis Minimal Lesion (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=251) | Testosterone (N=1019)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 8 (9)
Nausea (Gastrointestinal disorders) | 5 (5) | 10 (11)
Application Site Reaction (General disorders) | 47 (50) | 180 (196)
Nasopharyngitis (Infections and infestations) | 11 (12) | 22 (26)
Sinusitis (Infections and infestations) | 5 (5) | 25 (27)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (11) | 28 (32)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 24 (31)
Weight Increased (Investigations) | 5 (5) | 51 (51)
Headache (Nervous system disorders) | 8 (8) | 22 (26)
Depression (Psychiatric disorders) | 9 (10) | 13 (14)
Hirsutism (Skin and subcutaneous tissue disorders) | 4 (4) | 41 (48)
Hot Flush (Vascular disorders) | 5 (5) | 21 (21)
Hypertension (Vascular disorders) | 8 (8) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less